CLINICAL TRIAL: NCT01635140
Title: Prospective Randomized Trial of Hypofractionated Radiotherapy Versus Conventional Radiotherapy in Diffuse Brainstem Glioma in Children.
Brief Title: Hypofractionated Radiotherapy Versus Conventional Radiotherapy in Diffuse Brainstem Glioma in Children
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Children's Cancer Hospital Egypt 57357 (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CCHE-BT001
Record Dates: First submitted 2012-06-28; First posted 2012-07-09 (Estimated); Last update posted 2012-07-09 (Estimated); Status verified 2012-07

CONDITIONS: Pediatric Brain Stem Glioma
Keywords: DIPG; Hypofractionated Radiotherapy; Radiotherapy; Median survival
MeSH Terms: interventions — Radiation Dose Hypofractionation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Hypofractionated arm (Experimental): A total dose of 39 Gy in daily fractions of 3 Gy, 5 Fractions per week , by conformal radiotherapy sparing of the supratentorial brain. The planning target volume included the tumor as defined by the T2-weighted MRI images with a margin of 1.5-2.0 cm. Margins were adjusted for bony structures and tentorium. With exception of steroids, no neoadjuvant, concomitant, or adjuvant systemic treatment was allowed
  Interventions: Radiation: Hypofractionated radiotherapy
- Conventional arm (Other): The same planning and treatment procedures will be performed with the established conventional regimen: 54 Gy in 30 fractions giving 1.8 Gy per fraction.
  Interventions: Radiation: Conventional arm

INTERVENTIONS:
Radiation: Hypofractionated radiotherapy — A total dose of 39 Gy in daily fractions of 3 Gy, 5 Fractions per week
  Arms: Hypofractionated arm
Radiation: Conventional arm — A total dose of 54 Gy in 30 fractions giving 1.8 Gy per fraction.
  Arms: Conventional arm

SUMMARY:
Hypofractionated radiotherapy reduce the patient and family burden through decreasing the overall treatment time. This study is to evaluate the clinical end results of the hypofractionated radiotherapy in DIPG compared to the conventional treatment. The non-inferiority of the hypofractionated radiotherapy will result in decrease the hospital, stay or engagement, for more than its half with the same results.

DETAILED DESCRIPTION:
In lack of open study protocols aiming to increase cure rate in pediatric diffuse intrinsic pontine glioma (DIPG), the investigators examined a hypofractionated radiotherapy regimen up to a dose of 39Gy in 13 fractions, completed in 2.5-3 weeks, instead of 6 weeks.

This schedule offers a reduction in patient burden, especially preferable in children with a poor compliance and performance status. The non-inferiority of the hypofractionated regimen in its clinical end-results, with the reduction of the overall treatment time to less than its half will decrease the burden for the patient, his/her family and the treating department. This will be considered as added value without compromising the survival or increasing side effects.

ELIGIBILITY:
Inclusion Criteria:

1. Newly diagnosed patients with a diffuse intrinsic brainstem glioma, ages 3-18years, were eligible for this protocol.
2. Patients were required to have symptoms for less than 3 months and at least two findings of the neurologic triad: cranial nerve deficits, ataxia, or long tract signs.
3. No performance criteria were required for entry onto the study.
4. The diagnosis of DIPG based on a high-quality, gadolinium- enhanced magnetic resonance imaging (MRI) scan containing at least T1, T2 MRIs with gadolinium contrast in three series, as well as diffusion imaging.
5. Symptoms & signs of less than 3 months duration

Exclusion Criteria:

1. Children were not eligible if they had received any prior therapy other than steroid
2. The diagnosis of exophytic brainstem glioma

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 64 (Actual)
Dates: Start 2010-05; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Median overall-free survival | 3 years
Progression-free survival | 3 Years

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed s zaghloul, MD, Principal Investigator — Children's Cancer Hospital Egypt 57357
Locations (1):
- Children's Cancer Hospital Egypt 57357, Cairo, Egypt

REFERENCES:
- [Derived] Zaghloul MS, Eldebawy E, Ahmed S, Mousa AG, Amin A, Refaat A, Zaky I, Elkhateeb N, Sabry M. Hypofractionated conformal radiotherapy for pediatric diffuse intrinsic pontine glioma (DIPG): a randomized controlled trial. Radiother Oncol. 2014 Apr;111(1):35-40. doi: 10.1016/j.radonc.2014.01.013. Epub 2014 Feb 20. PMID 24560760